CLINICAL TRIAL: NCT03064893
Title: A Randomised Controlled Trial Comparing the Use of Alloderm Versus Dermacell in Immediate Implant Based Breast Reconstruction
Brief Title: The Use of Alloderm Versus Dermacell in Immediate Implant Based Breast Reconstruction
Acronym: REaCT-ADM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OTT 16-06
Record Dates: First submitted 2016-12-14; First posted 2017-02-27 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Breast Reconstruction
Keywords: acellular dermal matrix; mastectomy; breast reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dermacell (Active Comparator): Device for immediate implant based breast reconstruction
  Interventions: Device: Dermacell
- Alloderm (Active Comparator): Device for immediate implant based breast reconstruction
  Interventions: Device: Alloderm

INTERVENTIONS:
Device: Alloderm — Reconstruction material
  Arms: Alloderm
Device: Dermacell — Reconstruction material
  Arms: Dermacell

SUMMARY:
Breast reconstruction after mastectomy has been shown to provide psychosocial benefits to breast cancer patients and is considered an integral part of breast cancer treatment. In general, breast reconstruction can be accomplished using the patients own tissues or implantable prosthetic devices. Various acellular dermal matrices (ADMs) are offered on the market and the costs vary widely despite very similar qualities. The two most commonly used ADM products in North America by far are Dermacell and Alloderm. The difference between the two products include a) level of sterility, with Dermacell being sterilized to 10-9 while Alloderm is sterilized to 10-6 and b) the consistency and thickness of the biologic material and c) a significant different in cost ($2200 CAD vs $3600, respectively). Each product has shown to be safe and effective. As such, clinical equipoise exists. This will be a pragmatic trial to evaluate Dermacell with Alloderm in a head to head randomized fashion, with regards to the postoperative complications, namely infection, seroma formation (as measured by drain duration and output), loss of implant, incidence of revisional surgery and capsular contracture.

ELIGIBILITY:
Inclusion Criteria:

* Female patient
* Ages 20-90
* All patients undergoing mastectomy for breast cancer or prophylaxis for breast cancer with immediate implant-based reconstruction
* Able to provide verbal consent

Exclusion Criteria:

* Patients who have had prior chest wall or irradiation on the reconstructed side
* Patients not undergoing immediate breast reconstruction at the time of mastectomy
* Any patient with a contraindication to immediate breast reconstruction

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2019-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angel Arnaout, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arnaout A, Zhang J, Frank S, Momtazi M, Cordeiro E, Roberts A, Ghumman A, Fergusson D, Stober C, Pond G, Jeong A, Vandermeer L, Hutton B, Clemons M, On Behalf Of The REaCT Investigators. A Randomized Controlled Trial Comparing Alloderm-RTU with DermACELL in Immediate Subpectoral Implant-Based Breast Reconstruction. Curr Oncol. 2020 Dec 25;28(1):184-195. doi: 10.3390/curroncol28010020. PMID 33704185
- See also: The Rethinking Clinical Trials (REaCT) website — https://react.ohri.ca/

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: breasts
Period: Overall Study
Arm/Group | Dermacell | Alloderm
Started | 31; 40 breasts | 31; 41 breasts
Completed | 31; 40 breasts | 28; 38 breasts
Not Completed | 0; 0 breasts | 3; 3 breasts
Not completed — Change in surgery plan | 0 | 2
Not completed — Moved away | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dermacell | Alloderm | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: This is a baseline measure. The number of patients analyzed at baseline and follow-up are not equal.
  years | 51.4 (11.0) | 47.8 (11.1) | 49.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Female is an inclusion criteria.
  Participants
    Female | 31 | 31 | 62
    Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: This is a baseline measure. The number of patients analyzed at baseline and follow-up are not equal.
  participants
    Canada | 31 | 31 | 62
Smoking history [Count of Participants; unit: Participants] — Population: This is a baseline measure. The number of patients analyzed at baseline and follow-up are not equal.
  Participants
    Current | 1 | 3 | 4
    Prior (>1 or equal to month before) | 10 | 9 | 19
    Never | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Duration of Drain Placements
Description: Postoperative duration of drain placements for each postoperative breast.
Time Frame: within 6 months of initial surgery
Population: Participants may have had surgery on one or both breasts.
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: breasts
Arm/Group | Dermacell | Alloderm
Number analyzed (Participants) | 31 | 28
Number analyzed (breasts) | 40 | 38
days | 9.2 (4.5) | 10.8 (5.5)
Statistical Analysis 1: Comparison: Dermacell vs Alloderm; A minimum of 4 days between the two arms was considered clinically significant; Test type: Superiority; p = 0.15, t-test, 2 sided; Risk Difference (RD) = 1.6, 95% CI 2-sided [-0.7 to 3.9]

2. Secondary Outcome: Number of Breasts With an Episode of Seroma Formation Requiring Aspiration
Time Frame: within 6 months of initial surgery
Measure: Count of Units; unit: breasts
Units Other Than Participants: breasts
Arm/Group | Dermacell | Alloderm
Number analyzed (Participants) | 31 | 28
Number analyzed (breasts) | 40 | 38
breasts | 5 | 2

3. Secondary Outcome: Number of Breasts With Loss of Implant
Time Frame: within 6 months of initial surgery
Measure: Count of Units; unit: breasts
Units Other Than Participants: breasts
Arm/Group | Dermacell | Alloderm
Number analyzed (Participants) | 31 | 28
Number analyzed (breasts) | 40 | 38
breasts | 2 | 2

4. Secondary Outcome: Number of Breasts With Events of Revisional Surgery/ Return to Operating Room
Time Frame: within 6 months of initial surgery
Measure: Count of Units; unit: breasts
Units Other Than Participants: breasts
Arm/Group | Dermacell | Alloderm
Number analyzed (Participants) | 31 | 28
Number analyzed (breasts) | 40 | 38
breasts | 3 | 6

5. Secondary Outcome: Number of Breasts With Wound Dehiscence or Debridement
Description: Wound dehiscence is a post-operative complication. Wound debridement is a procedure. This outcome was collected on a post-surgery case report form.
Time Frame: within 6 months of initial surgery
Measure: Count of Units; unit: breasts
Units Other Than Participants: breasts
Arm/Group | Dermacell | Alloderm
Number analyzed (Participants) | 31 | 28
Number analyzed (breasts) | 40 | 38
breasts | 2 | 3

6. Secondary Outcome: Number of Breasts With Capsular Contracture (as Identified by the Plastic Surgeon)
Description: Capsular contracture is a post-operative complication identified by the plastic surgeon. This outcome was collected on a post-surgery case report form.
Time Frame: within 6 months of initial surgery
Measure: Count of Units; unit: breasts
Units Other Than Participants: breasts
Arm/Group | Dermacell | Alloderm
Number analyzed (Participants) | 31 | 28
Number analyzed (breasts) | 40 | 38
breasts | 0 | 1

7. Secondary Outcome: Number of Plastic Surgeon Visits
Time Frame: within 6 months of initial surgery
Population: The type of units is breasts. One participant could have had surgery on two breasts.
Measure: Median (Inter-Quartile Range); unit: visits
Units Other Than Participants: Breasts
Arm/Group | Dermacell | Alloderm
Number analyzed (Participants) | 31 | 31
Number analyzed (Breasts) | 40 | 38
visits | 3 [3 to 4.5] | 4 [3 to 5]

8. Secondary Outcome: Economics of Total Costs
Description: Economic impact will be assessed based on calculation of total costs with each material used to include the material costs, duration of operative room use, clinic and inpatient hospital costs, surgical billing costs and anaesthesia costs
Time Frame: 2 years
Population: Data for this outcome was not collected due to funding limitations. Data will not be collected in the future.
Arm/Group | Dermacell | Alloderm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was collected within 6 months of surgery (baseline).
Description: Serious adverse events and other adverse events collection/reporting were not reported. Adverse events were not included in the protocol as this was a pragmatic clinical trial comparing two standard of care interventions. Clinical complications were collected as secondary outcomes, which were collected by a variety study staff and not graded as adverse events (CTCAE).
Arm/Group | Dermacell | Alloderm
All-Cause Mortality (participants affected / at risk) | 1/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT03064893/Prot_SAP_000.pdf